CLINICAL TRIAL: NCT05906407
Title: COGNITION: Comprehensive Assessment of Clinical Features, Genomics and Further Molecular Markers to Identify Patients with Early Breast Cancer for Enrolment on Marker Driven Trials (Molecular Diagnostic Platform)
Brief Title: COGNITION: Genomics-Guided Precision Oncology in Early High-Risk Breast Cancer
Acronym: COGNITION
Status: Recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: S-790/2018; 01EK2202A (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung - BMBF)
Record Dates: First submitted 2022-12-08; First posted 2023-06-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Early-Stage Breast Cancer; Neoadjuvant Therapy
Keywords: Early Breast Cancer; Precision Oncology; Personalized Oncology; Genomic Profiling; Genomics-Guided Biomarker-Stratification; Postneoadjuvant-Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Profile; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh-frozen tissue and EDTA-blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Genomic Profiling / Sequencing — Procedure: genomic profiling (Whole-Genome- / Exome-Sequencing + RNA-Sequencing) in high-risk early breast cancer patients pre- and post neoadjuvant therapy

SUMMARY:
The COGNITION diagnostic platform elucidates the biomarker profile of neoadjuvant chemotherapy-resistant residual bulk tumors in high risk early breast cancer patients. The major goal is to provide a framework for genomic profiling, which serves as infrastructure for systematic biomarker-screening and -stratification for concise therapy-arm allocation in the interventional clinical phase II trial COGNITION-GUIDE (NCT05332561).

In patients, who display a poor response to standard-of-care neoadjuvant chemotherapy, tissue samples before and after neoadjuvant therapy are subjected together with blood samples to comprehensive genomic profiling to identify patients potentially benefiting from biomarker-guided interventions in COGNITION-GUIDE.

Samples not required for standard-of-care clinical procedures or genomic profiling are systematically collected in a dedicated bio-repository to fuel translational scientific companion programs. The continuously growing comprehensive database serves as an integrative resource for systematic, prospective multidimensional data collection (clinical records, biomaterial, genomic data).

In summary, the overarching goal is to generate a precision oncology platform i) to identify clinically-actionable biomarkers and drug targets that drive genomics-guided therapies and ii) to couple the observational, diagnostic registry platform to the independent, biomarker-stratified clinical therapy trial COGNITION-GUIDE.

DETAILED DESCRIPTION:
* Patient registration and enrolment: pts with histologically confirmed early breast cancer and indication for neoadjuvant chemotherapy (NACT, any subtype) who give their consent for the integrative genomic profiling study as pre-requisite for molecular stratification in the coupled phase II COGNITION-GUIDE (NCT05332561) therapy trial.
* Collection of biomaterial: Fresh-frozen tumor tissue from primary breast tumors is collected during routine procedures at study entry (T1: baseline-treatment naive) and from residual bulk tumors (T2: w/o pCR after NACT). To account for germline alterations (genomic control) and to fuel companion programs, consecutive blood samples are taken at baseline (V1) and after NACT (V2).
* Processing and analyses of patient samples: Biomaterials are centrally processed (standard histology/IHC and pathology review for tumor content; analyte extraction, QC according to standardized, quality-controlled, accredited workflows. Molecular profiling & clinical bioinformatics: Genomic profiling encompasses Whole-Genome on fresh-frozen tissue biopsies or Whole-Exome on FFPE surgical specimens (if fresh-frozen tissue has insufficient tumor cell content >20%). Both options are complemented by RNA-Seq facilitating an unbiased integrated view on the expression of multiple biomarkers.
* Clinical curation and data interpretation: Based on the curative intent, a rigorous, pre-defined biomarker algorithm (strong and soft biomarkers) is applied. This strategy allows assessment whether the tumor profile qualifies for one of the molecular-guided treatment arms.
* Molecular Tumor Board (MTB): Molecular data are interpreted by clinicians, bioinformaticians, molecular biologists, human geneticists and pathologists in a weekly interdisciplinary MTB established at NCT. Treatment-relevant biomarkers and actionable drug targets are validated independently. Disease-relevant germline alterations will lead to genetic counselling.
* Treatment recommendations and therapy implementation: Conclusive biomarker profiles from clinical, histopathological and genomic data drive assignment to one treatment arm. Therapeutic options are prioritized within a molecular report.
* Patient Monitoring / Follow-Up: Comprehensive documentation will be conducted at study entry and every 6 mths for 10 years.
* Pre-Clinical Companion Programs: The valuable pre- and post neoadjuvant biomaterial will be exploited to fuel collaborative studies around therapy failure, biomarker development and tracking of residual cancer burden in liquid biopsies (ctDNA).

ELIGIBILITY:
Inclusion Criteria:

* Female and male breast cancer patients aged ≥18 years.
* Patients with primary early breast cancer (irrespective of subtypes) or - as an exception - patients with isolated loco-regional relapses that can be treated with a curative intention
* Study entry is possible for patients with primary eBC at three timepoints:

  * Option A: patients planned to receive neoadjuvant chemotherapy are enrolled before starting the neoadjuvant treatment
  * Option B: patients with clinical non-complete response can be enrolled after the last cycle of neoadjuvant chemotherapy before surgery Note: Option A/B are strongly preferred entry time-points
  * Option C: eBC patients after surgery and planned or conducting standard-of-care (SoC) post-neoadjuvant chemotherapy can be enrolled after surgery until the last cycle of standard post-neoadjuvant chemotherapy, if they fulfill the following criteria

    * HER2+ BC or TNBC: non-pCR
    * HR+/HER2- BC: non-pCR and CPS-EG score ≥ 3 or non-pCR, ypN+ and CPS-EG-score ≥ 2 Note: Option C is not the preferred entry time-point Note: in case of loco-regional relapse, neoadjuvant treatment is not mandatory
* Patients must be willing to donate a recent tumour sample to the registry Note: fresh tumour tissue is preferred
* Patients, who agreed to and were able to sign the informed consent form (ICF).

Exclusion Criteria:

* Patients who did not sign or withdrew the informed consent form (ICF).
* Inability to retrieve tissue for molecular profiling Any physical or mental handicap or severe comorbidities that would hamper the adequate cooperation with the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk early-stage breast cancer (eBC) with suspected (non-clinical Complete Response - non-cCR ) and/or proven (non-pathological Complete Response - non-pCR) poor response towards NACT (irrespective of subtype).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive assessment of clinical patient data, collection of biomaterial and implementation of genomics- / molecular- and immune- guided precision medicine in eBC into the clinics. | 31/12/2028
  • Total number/percentage of patients with eBC and high risk for relapse i) eligible for genomic profiling, ii) successfully genomically-profiled tumours, iii) with conclusive biomarker profiles.
Setting up a clinical and multidimensional, molecular diagnostic registry platform for patients with eBC and high risk for relapse. | 31/12/2028
  • To record, show and benchmark the reality of high-throughput genomics-based medical care provided to patients with eBC and general outcome of patients (in terms of overall survival (OS), invasive disease-free survival (IDFS), distant disease-free survival (DDFS).
Assessment of feasibility and retrieval of the logistical, clinical and information basis to screen and enroll patients for independent molecular-driven intervention trials (independent of this registry, e.g. COGNITION-GUIDE). | 31/12/2028
  • Total number/percentage of patients enrolled in subsequent interventional trials.

SECONDARY OUTCOMES:
Identification and characterization of prognostic and predictive biomarkers, drug targets, resistance mechanisms and the immune environment. | 31/12/2028
  • Generation of catalogues of molecular aberrations, prognostic and predictive biomarkers and association between specific biomarkers and response to standard-of care treatment and/or targeted treatment for eBC (outside COGNITION) measured as OS, IDFS and DDFS.
Monitoring of treatment response and elucidation of resistance mechanisms using liquid biopsies. | 31/12/2028
  • Association between the detection of circulating tumour cells (CTCs), circulating tumour DNA (ctDNA) and outcome measured as OS, IDFS and DDFS.
Ex vivo cultivation of patient-derived biomaterial for research purposes. | 31/12/2028
  * Evaluation of the suitability of ex vivo model systems and liquid biopsy approaches (e.g. CTCs, ctDNA) to capture tumour heterogeneity, tumour-microenvironment interactions and drug response.
  * Characterization and modeling of the immune-compartment in tumour specimens and ex vivo culture approaches (immunoprofiling).
Delineation of tumour-microenvironment interactions with the immune systems. | 31/12/2028
  • Descriptive assessment of the impact of germline alterations on drug-response and toxicity (pharmacogenomics) by generation of a comprehensive catalogue of alterations in conjunction with administered therapies and toxicities.
Characterization of genetic alterations affecting drug metabolism (pharmacogenomics). | 31/12/2028
  • Assessment of the technical validation rate of somatic and germline alterations or further alterations in specific pathways by independent methods.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lichter, PhD, Principal Investigator — German Cancer Research Center (DKFZ) Heidelberg; Andreas Schneeweiss, MD, Principal Investigator — National Center for Tumor Diseases, Heidelberg; Verena Thewes, PhD, Principal Investigator — National Center for Tumor Diseases, Heidelberg
Locations (12):
- Germany (12):
  - University Hospital Augsburg, Augsburg
  - Charité - Berlin, Berlin
  - University Hospital Köln, Cologne
  - Medical Faculty and University Hospital Carl Gustav Carus, Dresden
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - National Center for Tumor Diseases (NCT) Heidelberg, Heidelberg
  - Caritas Hospital St. Josef, Regensburg
  - Robert Bosch Hospital Stuttgart, Stuttgart
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No